CLINICAL TRIAL: NCT01733615
Title: Discovering New Biomarkers for Monitoring Disease Progression in Patients With Mucopolysaccharidosis IVA (MPSIVA)
Brief Title: Discovering New Biomarkers For Monitoring Disease Progression in Patients With Mucopolysaccharidosis IVA
Status: Terminated | Type: Observational
Why Stopped: Original PI relocated to another institution
Sponsor: Emory University (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Madhuri Hegde, Associate Professor, Emory University
Other Study IDs: IRB00058450
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Mucopolysaccharidosis Type IVA
Keywords: Mucopolysaccharidosis Type IVA; Mucopolysaccharidosis Type IV; MPS Type IVA; MPS Type IV; Morquio Syndrome; Morquio Syndrome Type A; Urine biomarkers
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mucopolysaccharidosis IVA: Patients with the condition.

SUMMARY:
The purpose of this study is to find out more about some of the unusual chemicals (called oligosaccharides) that can occur naturally as a result of processes in the body. Researchers want to look at how these chemicals change with time and how they change between different patients with MPSIVA. These unusual chemicals were recently discovered in the urine from patients with MPSIVA. The investigators would like to study these chemicals before a specific enzyme replacement therapy is used. If the investigators understand how these chemicals change, the investigators may be able to use them to monitor this condition in the near future as well as help doctors know whether certain therapies work well in their patients.

DETAILED DESCRIPTION:
This is not a clinical trial and there is no outcome measurement. The biomarkers in this study are oligosaccharides that secreted in the urine from patients with MPSIVa. In this study, we will try to define the variability of these oligosaccharides in the same patient at different time points, including different month of a year and different collections during the day as well as variations of these oligosaccharide in different affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mucopolysaccharidosis IVA

Exclusion Criteria:

* Patients receiving enzyme replacement therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed or untreated Mucopolysaccharidosis IVA patients across the nation collected from national major genetic laboratories, national major genetic clinics, Includes the Emory Genetics Clinic, Mayo Clinic, UPMC, Children's Hospital of Philadelphia, and Nationwide Children's Center in Washington, DC.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Quantification of urinary oligosaccharides in urine from a first morning void in patients with Mucopolysaccharidosis IVA. | Every 2 months over the course of a year.
  The variability of oligosaccharides in the same patient over different time points and urine specimen type will be evaluated.

SECONDARY OUTCOMES:
Quantification of urinary oligosaccharides in urine from a random collection in patients with Mucopolysaccharidosis IVA. | One urine over the course of a year or 6M
  The variability of oligosaccharides among different patients with MPSIVa will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Madhuri Hegde, PhD, FACMG, Principal Investigator — Emory University
Locations (1):
- Emory University, Dept of Human Genetics, Decatur, Georgia, United States

REFERENCES:
- [Background] Tiede S, Storch S, Lubke T, Henrissat B, Bargal R, Raas-Rothschild A, Braulke T. Mucolipidosis II is caused by mutations in GNPTA encoding the alpha/beta GlcNAc-1-phosphotransferase. Nat Med. 2005 Oct;11(10):1109-12. doi: 10.1038/nm1305. Epub 2005 Oct 2. PMID 16200072
- [Background] Walkley SU, Thrall MA, Haskins ME, Mitchell TW, Wenger DA, Brown DE, Dial S, Seim H. Abnormal neuronal metabolism and storage in mucopolysaccharidosis type VI (Maroteaux-Lamy) disease. Neuropathol Appl Neurobiol. 2005 Oct;31(5):536-44. doi: 10.1111/j.1365-2990.2005.00675.x. PMID 16150124